CLINICAL TRIAL: NCT05161026
Title: Impact of Allo-HSCT on Bone Remodeling: Evolution of Bone Mineral Density and Architecture Measured by Bone Densitometry Coupled With FRAX / TBS in Allo-HSCT
Brief Title: Impact of Allo-HSCT on Bone Remodeling: Evolution of Bone Mineral Density and Architecture Measured by Bone Densitometry
Acronym: REMODALLO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-047
Record Dates: First submitted 2021-07-13; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Myeloid Leukemia, Acute
Keywords: allo-HSCTs transplant; osteoporosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with AML (Other): Patients with AML
  Interventions: Other: Bone osteodensitometry

INTERVENTIONS:
Other: Bone osteodensitometry — Evaluation of bone osteodensitometry

SUMMARY:
Evaluation of variation of mineral density and bone microarchitecture after allogeneic HSCTs transplant in hematologic malignancies. Comparison with the general population.

DETAILED DESCRIPTION:
Allo-HSCTs performed for the treatment of hematologic malignancies has been increasing in recent years. There is therefore a growing interest in the quality of life of these patients and in particular for the bone complications of the transplant. Indeed, it was found a high incidence of osteoporosis / osteopenia in this population associated with an increased risk of osteoporotic fracture from 6 to 9 times compared to the general population.

This study will evaluate the variation of mineral density and bone microarchitecture parameters by bone densitometry with measurement of trabecular bone score and fracturing risk before and after allogeneic HSCTs transplant, at predefined times. It's also evaluating pain scale, fracture incidence and bone remodeling markers.

ELIGIBILITY:
Inclusion Criteria:

* Cytological diagnosis of acute myeloid leukemia (AML) with indication for a first-line allo-HSCTs transplant
* Patient affiliated to the social security system
* For women of childbearing age, use of reliable contraception throughout the study in accordance with the CPR of the drugs used.
* The patient must be able to comply with study visits and per protocol procedures
* Patient who has been informed of the study and has signed his informed consent

Exclusion Criteria:

* Person under guardianship or curatorship, or unable to understand the purpose of the study.
* Hematologic malignancies other than AML
* History of neoplasia with bone involvement (sarcoma, multiple myeloma, metastasis...) and/or any solid cancer less than 5 years old
* History of fracture of the femoral neck prior to the diagnosis of hematologic malignancies
* Known bone involvement related to AML at diagnosis
* Primary or secondary osteoporosis known to the diagnosis of hematologic malignancies
* Corticotherapy > 3 months at a dose > 7.5mg/day prior to the diagnosis of hematological disease
* Autograft or anterior allograft
* Pathologies influencing bone metabolism: known inflammatory rheumatism (rheumatoid arthritis, ...), primary hyperparathyroidism, chronic renal failure (GFR < or = at 30ml / min / 1.73m2)
* Pregnant or lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
bone mineral density evaluation | change over time between diagnostic, transplant, 6 months and 12 months post-transplant
  bone mineral density evaluation post-transplant

SECONDARY OUTCOMES:
bone mineral density evaluation | change over time between 24 months and 36 months post-transplant
  long term bone mineral density evaluation
Bone architectural abnormalities and fracture risk | change over time between diagnostic, transplant, 6 months and 12 months post-transplant
  evaluation of bone architectural abnormalities and fracture risk
bone remodeling markers | change over time between diagnostic, transplant, 6 months and 12 months post-transplant
  Dosage of bone remodeling markers
Pain evaluation | change over time between diagnostic, transplant, 6 months, 12 months, 24 months and 36 months post-transplant
  Pain evaluation (EVA)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Amiens, Amiens
  - CHU CAEN, Caen
  - Chu Lille, Lille
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No